CLINICAL TRIAL: NCT00683722
Title: A Phase II, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of PROCHYMAL™ (ex Vivo Cultured Adult Human Mesenchymal Stem Cells) Intravenous Infusion for the Treatment of Subjects With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: PROCHYMAL™ (Human Adult Stem Cells) for the Treatment of Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mesoblast, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 801
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Pulmonary Emphysema; Chronic Bronchitis
Keywords: COPD; Airflow Obstruction, Chronic; Chronic Airflow Obstruction; Chronic Obstructive Airway Disease; Chronic Obstructive Lung Disease; Chronic Obstructive Pulmonary Disease; Pulmonary Emphysema; Chronic Bronchitis; Mesenchymal Stem Cells (MSCs); Adult Human Stem Cells; Osiris; Prochymal™
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Emphysema; Bronchitis, Chronic | interventions — remestemcel-l

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prochymal™ (Experimental): Participants received Prochymal™ a total of 400×10^6 cells, intravenous (IV) infusions on Days 0, 30, 60, and 90.
  Interventions: Drug: Prochymal™
- Placebo (Placebo Comparator): Participants received placebo-matching IV infusions on Days 0, 30, 60 and 90.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prochymal™ — IV infusion of ex- vivo cultured adult human mesenchymal stem cells.
  Arms: Prochymal™
Drug: Placebo — IV infusion of excipient of Prochymal™.
  Arms: Placebo

SUMMARY:
The objective of the present study is to establish the safety and efficacy of multiple administrations of Prochymal™(ex-vivo cultured human adult mesenchymal stem cells) in participants with moderate to severe chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
COPD is currently the fourth leading cause of death in the United States. It is clear that there is a significant unmet medical need for safe and effective therapies to treat moderate to severe COPD. This patient population has a high mortality rate and requires frequent hospitalizations due to disease-related exacerbations. Based on severity distribution estimates, approximately 70% of all current COPD patient have either moderate or severe COPD. COPD has no known cure, thus current therapeutic intervention is aimed at providing relief of symptoms. Oxygen therapy is the only treatment that has been shown to improve survival. Smoking cessation has been shown to slow the rate of forced expiratory volume in 1 second (FEV1) decline and COPD progression. In general patient are treated with bronchodilators and inhaled corticosteroids, but again, these measures do not provide any significant benefit regarding disease progression or prognosis. The characteristics and biologic activity of Prochymal™, along with a good safety profile in human trials to date, suggest that Prochymal™ may be a good candidate for addressing this unmet medical need.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a diagnosis of moderate or severe COPD.
* Participant must have a post-bronchodilator FEV1/forced vital capacity (FVC) ratio < 0.7.
* Participant must have a post-bronchodilator FEV1 % predicted value ≥ 30% and < 70%.
* Participant must be between 40 and 80 years of age, of either sex, and of any race.
* Participant must be a current or ex-smoker, with a cigarette smoking history of ≥ 10 years or > 10 pack-years.

Exclusion Criteria:

* Participant has been diagnosed with asthma or other clinically relevant lung disease other than COPD (e.g. restrictive lung diseases, sarcoidosis, tuberculosis, idiopathic pulmonary fibrosis, bronchiectasis, or lung cancer).
* Participant has been diagnosed with α1-antitrypsin deficiency.
* Participant has a body mass greater than 150 kg (330 lb) or less than 40 kg (88 lb).
* Participant has active infection.
* Participant has had a significant exacerbation of COPD or has required mechanical ventilation within 4 weeks of screening.
* The participant with clinically relevant uncontrolled medical condition not associated with COPD.
* Participant has documented history of uncontrolled heart failure.
* Participant has pulmonary hypertension due to left heart condition.
* Participant has atrial fibrillation or significant congenital heart defect/disease.
* Participant has initiated pulmonary rehabilitation within 3 months of screening.
* Participant is allergic to bovine or porcine products.
* Participant has evidence of active malignancy, or prior history of active malignancy that has not been in remission for at least 5 years.
* Participant has a life expectancy of < 6 months.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-03-20 (Actual); Primary Completion 2009-03-09 (Actual); Study Completion 2010-08-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 2 Years

SECONDARY OUTCOMES:
Change from Baseline in Pulmonary Function Test: Forced Expiratory Volume (FEV)1 at Year 1 and Year 2 | Baseline, Year 1, Year 2
Change from Baseline in Pulmonary Function Test: Forced Expiratory Volume (FEV)1 %predicted at Year 1 and Year 2 | Baseline, Year 1, Year 2
Change from Baseline in Pulmonary Function Test: Forced Vital Capacity (FVC) at Year 1 and Year 2 | Baseline, Year 1, Year 2
Change from Baseline in Pulmonary Function Test: Forced Vital Capacity (FVC) %predicted at Year 1 and Year 2 | Baseline, Year 1, Year 2
Change from Baseline in Pulmonary Function Test: Forced Expiratory Volume to Forced Vital Capacity Ratio (FEV1/FVC) at Year 1 and Year 2 | Baseline, Year 1, Year 2
Change from Baseline in Diffusing capacity of the lung for carbon monoxide (DLCO) at Year 1 and Year 2 | Baseline, Year 1, Year 2
Change from Baseline in Diffusing capacity of the lung for carbon monoxide (DLCO) %predicted at Year 1 and Year 2 | Baseline, Year 1, Year 2
Change from Baseline in Alveolar Volume (VA) at Year 1 and Year 2 | Baseline, Year 1, Year 2
Change from Baseline in Diffusing capacity of the lung for carbon monoxide to Alveolar Volume ratio (DLCO/VA)at Year 1 and Year 2 | Baseline, Year 1, Year 2
Change from Baseline in Functional residual capacity (FRC) at Month 6 | Baseline, Month 6
Change from Baseline in Total Lung Capacity (TLC) at Month 6 | Baseline, Month 6
Change from Baseline in Residual Volume (RV) at Month 6 | Baseline, Month 6
Change from Baseline in Airway Resistance (RAW) at Month 6 | Baseline, Month 6
Change from Baseline in 6-Minute Walk Test at Year 1 and Year 2 | Baseline, Year 1, Year 2
  Change from baseline in the total distance walked in 6 minutes was reported.
Change from Baseline in Borg Dyspnea Scale at Year 2 | Baseline, Year 2
Change from Baseline in Health-related quality of life: St George's Respiratory Questionnaire (SGRQ) at Year 1 and Year 2 | Baseline, Year 1, Year 2
Change from Baseline in Physician Global Assessment Scale at Year 1 and Year 2 | Baseline, Year 1, Year 2
  The physician evaluated the subject's global status as improved, unchanged, or worsened from pretreatment.
Time to COPD Exacerbation | Up to 2 Years
Number of COPD Exacerbations | Up to 2 Years
Change from Baseline in Pulmonary Hypertension at Month 6 | Baseline, Month 6
Change from Baseline in Systemic Inflammation at Year 1 and Year 2 | Baseline, Year 1 and Year 2
  Changes in systemic inflammation was determined by C-Reactive Protein (CRP) assays.

CONTACTS AND LOCATIONS:
Overall Officials: Mahboob Rahman, MD, Study Director — Mesoblast, Inc.
Locations (6):
- United States (6):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Los Angeles Biomedical Research Institute at Harbor UCLA Medical Center, Torrance, California
  - American Health Research, Charlotte, North Carolina
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Vermont Lung Center, University of Vermont, Burlington, Vermont

REFERENCES:
- [Derived] Weiss DJ, Segal K, Casaburi R, Hayes J, Tashkin D. Effect of mesenchymal stromal cell infusions on lung function in COPD patients with high CRP levels. Respir Res. 2021 May 8;22(1):142. doi: 10.1186/s12931-021-01734-8. PMID 33964910
- [Derived] Weiss DJ, Casaburi R, Flannery R, LeRoux-Williams M, Tashkin DP. A placebo-controlled, randomized trial of mesenchymal stem cells in COPD. Chest. 2013 Jun;143(6):1590-1598. doi: 10.1378/chest.12-2094. PMID 23172272
- [Derived] Gross NJ. The COPD Pipeline XIV. COPD. 2012 Feb;9(1):81-3. doi: 10.3109/15412555.2012.646587. No abstract available. PMID 22292600